CLINICAL TRIAL: NCT02051829
Title: Comparison of Preoperative Screening Score for OSA
Brief Title: Comparison of Preoperative Screening Score for Obstructive Sleep Apnea (OSA)
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, FCCP, Eric DEFLANDRE, MD, FCCP, Astes
Other Study IDs: SEED-ASTES-2014
Record Dates: First submitted 2014-01-24; First posted 2014-01-31 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: Comparison of the four screening score
  Interventions: Other: Comparison of the four screening score

INTERVENTIONS:
Other: Comparison of the four screening score — Comparison of the four screening score, for patient making a preoperative assessment for SLBO (clinique Saint-Luc de BOuge)

SUMMARY:
Comparison of preoperative screening score for OSA. In a preoperative population, comparison of the STOP-BANG, DES-OSA, P-SAP and OSA50 score.

DETAILED DESCRIPTION:
Comparison of preoperative screening score for OSA (Obstructive Sleep Apnea). In a preoperative population, comparison of the STOP-BANG, DES-OSA, P-SAP and OSA50 score.

Comparison between scores and if applied with the results of a polysomnography (PSG).

ELIGIBILITY:
Inclusion Criteria:

* All adults patients (> 18 years) performing a preoperative assessment at the ASTES Doctor's Office (ASTES is an acronym with the name of Medical Doctors involved in this office)

Exclusion Criteria:

* Patients < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (> 18 years) presenting for preoperative assessment before surgery at SLBO.
Sampling Method: Non-Probability Sample
Enrollment: 1584 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with a positive DES-OSA score | Baseline
  Comparison of the result of the DES-OSA score with results of previously describes scores (STOP-BANG, OSA50 and P-SAP).

SECONDARY OUTCOMES:
Number of patients with a positive STOP-Bang score and a positive PSG (PolySomnoGraphy) | Baseline
  For the patients with a positive STOP-Bang score: we will make a PSG. After this one, we will compare the result of four scores (STOP-Bang, OSA50, P-SAP and DES-OSA) and the result of the PSG (especially AHI: Apnea Hypopnea Index)

CONTACTS AND LOCATIONS:
Overall Officials: Eric P DEFLANDRE, MD, FCCP, Principal Investigator — Astes
Locations (1):
- Cabinet Medical ASTES, Jambes, Jambes, Belgium

REFERENCES:
- [Derived] Deflandre E, Degey S, Brichant JF, Donneau AF, Frognier R, Poirrier R, Bonhomme V. Pre-Operative Ability of Clinical Scores to Predict Obstructive Sleep Apnea (OSA) Severity in Susceptible Surgical Patients. Obes Surg. 2017 Mar;27(3):716-729. doi: 10.1007/s11695-016-2352-4. PMID 27599985